CLINICAL TRIAL: NCT00428831
Title: Clinical Correlates to Influenza Genomic Data
Brief Title: Clinical IGSP-CHOP Boston
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06-0096
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2008-09

CONDITIONS: Influenza
Keywords: influenza, genomic data, nasopharyngeal aspirate
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients with respiratory illnesses.

SUMMARY:
The main purpose of this study is to look at relationships between types of flu viruses and characteristics of infected patients, including vaccination status, organ system involvement, and disease severity. In this study, 500 patients with respiratory illnesses will have nose/throat fluid samples collected. At Children's Hospital Boston, patients 30 days to 5 years of age will be recruited; at Beth Israel Deaconess Medical Center, patients of any age will be eligible. The researchers will compare the symptoms of infection by similar flu virus types and look at differences in the flu virus types between the 2 age groups of patients. The researchers will also look at whether any flu virus types first show up in the children prior to infecting the adults. Hopefully this study will improve understanding of how flu viruses develop, spread, and cause disease. This information may help the development of more effective flu vaccines, prevention measures, and treatments.

DETAILED DESCRIPTION:
There is evidence that the pediatric population, in particular, may play an essential role in influenza transmission. One recent study showed that children between the ages of 3 and 4 years were consistently the first population group to be affected by influenza illness over several winter seasons. In addition, influenza illness in children less than 5 years of age was the strongest predictor of mortality among adults. Collecting samples from adults as well as children in the pre-school age group would enable researchers to further examine the specific role this population plays in the evolution of influenza virus lineages and the development of dominant strains. In this prospective observational study, the researchers are therefore proposing to collect samples from pediatric patients at Children's Hospital and from adults at Beth Israel Deaconess Medical Center. This will enable the researchers to compare the clinical manifestations resulting from infection by similar strains and to examine differences in the genomic sequences of the viruses between the two population groups. The primary objective of this study is to conduct a pilot study to explore correlations between influenza viral strains and clinical characteristics of infected patients, including vaccination status, organ system involvement, and disease severity. With regard to outcome measures, the researchers will determine rates of clinical features associated with specific viral strains. The clinical characteristics the researchers will examine are vaccination status, illness symptoms (presence of fever, cough, runny nose/ stuffy nose, headache, myalgia, fatigue), initial O2 saturation, treatment with antibiotics or antivirals, hospitalization, daycare or kindergarten attendance, exposure to elderly persons, and length of illness. The secondary study objective is to conduct a pilot study to compare the influenza genomic sequences and clinical data from pediatric and adult patients infected with influenza and to explore potential viral transmission patterns between these two populations. With regard to the outcome measures, the researchers will determine rates of clinical features and of specific viral strains in the pediatric and adult populations. The clinical characteristics the researchers will examine are the same as in the primary objective. The researchers will also identify any temporal patterns in the infections caused by specific viral strains in the two groups. Specifically, the researchers will examine whether any viral strains first emerge in the pediatric population prior to infecting the adult group. A total of 500 patients with respiratory illnesses will be recruited at Children's Hospital Boston and at Beth Israel Deaconess Medical Center. At Children's Hospital, patients 30 days to 5 years of age will be recruited; at Beth Israel Deaconess Medical Center patients of any age will be eligible. The researchers will recruit patients of both genders and of any health status. Respiratory samples and clinical information will be collected from each participant. It is hoped that this study will help further the researchers' understanding of how influenza viruses evolve, spread, and cause disease. In the future, this may help in the development of more effective vaccines and prevention measures, as well as treatments for people infected with influenza.

ELIGIBILITY:
Inclusion Criteria:

1. For pediatric population: Age of patient: 30 days - 5 years; for adult population: any age
2. Illness onset within past 5 days
3. Symptoms of fever (>=38°) plus one or more of the following: cough, runny nose, congestion, or sneezing (twice or more within one day). These symptoms must be present at the time of presentation to the emergency department (ED) or admission to the hospital.
4. Patient or parent/guardian is able to give informed consent

Exclusion Criteria:

1. Pediatric patient or non-verbal adult is not accompanied by a caregiver
2. Participant/caregiver cannot be reached by phone in 7-10 days
3. Patient has a condition that can compromise respiratory function or the handling of respiratory secretions (e.g., severe cognitive dysfunction, spinal cord injuries, or other neuromuscular disorders)

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Will recruit patients of both genders and of any health status. Will be recruited at Children's Hospital Boston and at Beth Israel Deaconess Medical Center. At Children's Hospital, patients 30 days to 5 years of age will be recruited; at Beth Israel Deaconess Medical Center patients of any age will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Patient's length of illness, symptoms, medication use, influenza vaccination status, initial O2 saturation, hospitalization, daycare or kindergarten attendance, exposure to elderly persons, and length of illness. | Enrollment and Follow up phone call.

SECONDARY OUTCOMES:
Rates of clinical features and of specific viral strains in the pediatric and adult populations. | Enrollment and Follow up phone call.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Boston - Infectious Diseases, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Medicine - Infectious Disease, Boston, Massachusetts